CLINICAL TRIAL: NCT01682499
Title: Calcium and Magnesium Infusion for the Prevention of Taxane Induced Neuropathy in Earlier Stage Breast Cancer
Brief Title: Calcium and Magnesium Infusion for the Prevention of Taxane Induced Neuropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB/COSA # 079-12
Record Dates: First submitted 2012-08-21; First posted 2012-09-11 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Paclitaxel-induced Neuropathy
Keywords: neuropathy; taxane; paclitaxel; calcium; magnesium; prevention
MeSH Terms: interventions — Calcium Gluconate; Magnesium Sulfate; Calcium; Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Calcium and Magnesium Infusion (Experimental)
  Interventions: Drug: calcium gluconate and magnesium sulfate

INTERVENTIONS:
Drug: calcium gluconate and magnesium sulfate — Intravenous calcium gluconate and magnesium sulfate, 1g each agent in 100 ml D5W over 30 minutes, immediately before and after each dose of paclitaxel
  Other Names: Ca; Mg; Calcium; Magnesium

SUMMARY:
This is a pilot study evaluating the feasibility of intravenous calcium and magnesium (Ca/Mg) infusion for prevention of taxane induced neuropathy in patients with early stage breast cancer receiving adjuvant or neo-adjuvant paclitaxel, either given every 2 weeks for 4 cycles or every week for 12 weeks.

DETAILED DESCRIPTION:
Chemotherapy induced peripheral neuropathy (CIPN) is a major dose limiting side effect of many cytotoxic chemotherapy, and can be extremely disabling, causing significant loss of functional abilities. Calcium and magnesium infusions were shown to decreased the incidence and intensity of neuropathy symptoms related to oxaliplatin.

There are currently no effective drugs or treatment modalities for the prevention or treatment of taxane related neuropathy. Given the morbidity of taxane induced neuropathy and the safety of Ca/Mg infusion, it is reasonable to assess the feasibility of this intervention in woman with stage I-III breast cancer receiving adjuvant or neo-adjuvant paclitaxel treatment, either given every 2 weeks for 4 cycles or every week for 12 weeks. Calcium gluconate and magnesium sulfate, 1 g of each agent in 100 ml D5W will be infused over 30 minutes, immediately before and after each dose of paclitaxel. The Ca/Mg infusion will be given through the same line used for giving chemotherapy.

The primary aim of this study is to assess paclitaxel-related neuropathy (grade 2 or greater) as measured by NCI Common Terminology Criteria Version 3 in patients receiving Ca/Mg infusion during paclitaxel chemotherapy and compare it with historical controls. Secondary endpoints will include other measures of neuropathy and quality of life such as the FACT-Tax score, taxane-related neuropathy pain as measured by the Brief Pain Inventory-Short Form (BPI-SF), and measure of cognitive impairment using FACT-cog score.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* History of stage I-III breast cancer
* Patient scheduled to be receiving adjuvant or neo-adjuvant paclitaxel given every week for 12 weeks or given every two weeks for 4 cycles
* Serum magnesium level ≤ UNL
* Serum calcium level ≤ UNL
* Serum creatinine ≤ 1.5 x UNL
* Signed informed consent

Exclusion Criteria:

* Pre-existing peripheral neuropathy of any grade
* Current treatment for arrhythmias
* Concurrent treatment with anticonvulsants, tricyclic antidepressants, or other neuropathic medications such as carbamazepine, phenytoin, gabapentin, lamotrigine, or concurrent treatment with other neuropathic chemotherapy agents
* Current narcotic use

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
to assess paclitaxel-related neuropathy (grade 2 or greater) | 2 years
  The primary aim of this study is to assess paclitaxel-related neuropathy (grade 2 or greater) as measured by NCI Common Terminology Criteria Version 3 in patients receiving Ca/Mg infusion during paclitaxel chemotherapy and compare it with historical controls

SECONDARY OUTCOMES:
Other measures of neuropathy and quality of life | 2 years
  The secondary endpoints will include other measures of neuropathy and quality of life such as the FACT-TAX score
Taxane-related neuropathic pain | 2 years
  Taxane-related neuropathic pain as measured by the Brief Pain Inventory-Short Form (BPI-SF)
Measure of cognitive impairment | 2 years
  Measurement of cognitive impairment using FACT-Cog score

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Shao, MD, Principal Investigator — Beth Israel Medical Center
Locations (3):
- United States (3):
  - Beth Israel Medical Center, New York, New York
  - Beth Israel Comprehensive Cancer Center, New York, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York